CLINICAL TRIAL: NCT03307356
Title: The University of Pennsylvania Uterus Transplant for Uterine Factor Infertility Trial
Acronym: UNTIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 827853
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome; Uterine Agenesis; Infertility, Female, of Uterine Origin; Uterine Factor Infertility
Keywords: Uterine Transplant; MRKH
MeSH Terms: conditions — Mullerian aplasia; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterine Transplantation (Experimental): Women will undergo extensive medical and psychological screening. Five women that meet all inclusion and exclusion criteria will undergo ovarian stimulation, oocyte retrieval and will create embryos that will be stored for future use. Women will then undergo uterine transplantation from a donor. Following transplant women will be closely monitored for complications (including infection and rejection). If no complications arise, or complications that do arise can be treated, attempts at pregnancy will begin approximately 6 months after transplant. Pregnancy in the setting of uterine transplant requires directly placing embryos directly into the uterus.
  Interventions: Other: Uterine Transplant

INTERVENTIONS:
Other: Uterine Transplant — Transplant of a uterus from a donor, deceased or living
  Other Names: Donor Uterine Transplant

SUMMARY:
Options for childbearing are limited for the thousands of women in the United States who suffer from absolute uterine factor infertility. Uterine transplantation is an emerging treatment that provides hope for these individuals.

In the Penn UNTIL trial, the investigators plan to perform uterus transplants on five women who will ultimately undergo embryo transfer, pregnancy, delivery, and then transplant hysterectomy.

This trial is accepting women in need of a transplant and also women who are interested in being a live donor.

For more information please visit: https://clinicalresearch.itmat.upenn.edu/clinicaltrial/4821/congenital-abnormalitiesfemale-infertility-penn-ut/

DETAILED DESCRIPTION:
BACKGROUND The inability to conceive children can be one of the most devastating and traumatic situations to arise in the life of an individual or couple. While assisted reproductive technologies have been developed that help overcome many causes of infertility, uterine factor infertility has remained an intractable condition. Absolute uterine factor infertility (AUFI) occurs when the uterus is either not present (congenitally absent or surgically removed) or is present but is not capable of sustaining a pregnancy. AUFI can result from either congenital absence of a uterus (Mayer-Rokitansky-Kuster-Hauser [MRKH] syndrome) or other Müllerian anomalies. MRKH occurs in 1:4000 of females. It is difficult to determine the exact number of women that suffer from AUFI, however estimates are as high as 7 million women between the ages of 15-34 may suffer from this condition in the United States.

Existing options for individuals with AUFI to achieve parenthood are adoption and the use of a gestational carrier. Use of a gestational carrier is the only alternative that allows an individual or couple to have a child genetically related to the intended parent(s). These options are considered acceptable to many women with AUFI; however, there are a number of significant limitations to these alternatives. The use of a gestational carrier is fraught with ethical, legal, and social controversy because it shifts the burden of gestation from one woman to another, usually for payment. Additionally, adoption and/or surrogacy may not be permissible to a couple due to social, ethical, moral or religious considerations. If these alternatives are acceptable to a couple, they may not be affordable. Finally, these alternatives may not be accessible as barriers to domestic and international adoption have increased and the use of a compensated gestational carrier is not legally protected in most states (and is illegal in some states). The limitations of these alternatives may account for the extraordinary interest in UTx by women with AUFI, as 92% of women with AUFI would undergo UTx as first line management for their AUFI, above adoption and surrogacy.

Understanding the limitations of these alternatives, uterine transplantation (UTx) began to be explored as a concept in animal studies in the 1970s. In 2012, a Swedish team led by Dr. Mats Brannstrom started the first human uterine transplantation trial. The first live birth after successful UTx occurred in Sweden in 2014. As of September 2021, the investigators estimate 33 uterus transplants have been performed in the United States and >10 babies have been born to these women.

Unlike all other transplants, uterine transplantation is "ephemeral". This means that a uterine transplant is only maintained during the individual's child-bearing period which, in the case of uterine transplantation, will be the time necessary to produce one or two children (<10 years). Although pregnancy after transplant is considered high risk, more than 15,000 babies have been born to female recipients of solid organ transplants that were immunosuppressed with no reported increased risk of fetal malformations.

STUDY DESIGN Recognizing that the University of Pennsylvania has been a leader in all of the domains required to build a successful uterus transplant program, planning for the Penn UNTIL trial began in October 2016. The UNTIL trial is is a nonrandomized, interventional human study whose goal is to achieve live birth after donor uterus transplantation. The investigators plan to perform approximately five uterus transplants in this pilot trial. Prior to being listed for transplant, the participants will need to create embryos through ovarian stimulation, oocyte retrieval and in vitro fertilization that will be cryopreserved. After undergoing donor uterus transplantation, participants will be monitored for rejection, infection and other complications for twelve months.

If the graft is clinically stable and any complications that arise are successfully treated 6 months after transplantation, the embryos created prior to transplantation will be directly placed into the uterus in order for the women to achieve pregnancy. If pregnancy is achieved the participant will be monitored by a Maternal Fetal Medicine specialist (high-risk obstetrician) with goal to deliver at 37-39 weeks unless otherwise indicated. All deliveries will occur via cesarean delivery. If the participant and partner wish to attempt an additional pregnancy and the medical team feel it is safe to proceed, attempts at a second pregnancy will be undertaken. Again, if pregnancy is achieved following embryo transfer the participant will be monitored for the duration of her pregnancy by a Maternal Fetal Medicine specialist with goal to deliver at 37-39 weeks through repeat cesarean delivery unless otherwise indicated. Hysterectomy will either be performed at the time of cesarean delivery or shortly following the final cesarean delivery.

The transplanted uteri will be from either living or deceased donors. Interested potential donors will be screened and evaluated and if eligible with continued interest in participation, will undergo radical hysterectomy for the purpose of uterus transplant into a woman with AUFI. Deceased donors will be considered and screened with the organ procurement organization Gift of Life Donation Program.

For more information please visit: https://clinicalresearch.itmat.upenn.edu/clinicaltrial/4821/congenital-abnormalitiesfemale-infertility-penn-ut/

ELIGIBILITY:
Uterine Transplant Recipient Participant Inclusion Criteria:

1. XX-bearing individual diagnosed with Uterine Factor Infertility (UFI) a
2. Age 21-40
3. Lives in Philadelphia region for the duration of the trial
4. Received counseling regarding alternatives to uterine transplant such as adoption or surrogacy
5. Intact ovaries
6. Vaginal length >6 cm (average vaginal length established with dilators)
7. Body mass index <35 kg/m2
8. Fluent in the English Language
9. If cervix present/previously present, human papillomavirus (HPV)) negative or received vaccination for HPV
10. Willing to comply with screening, protocol and all required procedures
11. Has adequate social support
12. Has undergone controlled ovarian hyperstimulation, egg retrieval, in vitro fertilization, and embryo freezing and has frozen embryos of sufficient embryo quality/quantity (≥2 high quality blastocysts); (Required for Transplant Phase, not Screening or Evaluation Phases)

Uterine Transplant Recipient Participant Exclusion Criteria:

1. Previous multiple major abdominal/pelvic surgery
2. Severe endometriosis
3. History of hypertension, diabetes mellitus, thrombophilia or other clotting or bleeding disorders, significant heart, liver, kidney or central nervous system disease
4. History of prior malignancy except for cervical cancer in stage 1a or 1b (must be in remission for 3 years)
5. History of significant psychiatric illness
6. Allergy, hypersensitivity, or intolerance of expected immunosuppressive agents (i.e. Thymoglobulin®, tacrolimus, etc.)
7. Allergy, hypersensitivity, or intolerance of heparin or aspirin
8. Presence of active documented systemic infection or recent systemic infection within the past 3 months
9. Seropositivity for HIV, HBV core antibody or antigen, HCV
10. Current smoker (smoking cessation must have occurred 3 months prior to enrollment)
11. Chemical and/or alcohol dependency or abuse
12. Psychosocial problems (including alcoholism, drug abuse, documented behavioral disorders)
13. Renal abnormalities, specifically single kidney or pelvic kidneys (imaging confirmation of 2 normal kidneys is required for MRKH subjects)
14. Contraindications to pregnancy
15. Unwilling to receive a transfusion of blood or blood products

Living Donor Participant Inclusion Criteria:

1. Age 30-50
2. Has definitively completed childbearing
3. Live birth to miscarriage ratio ≥1
4. Body mass index <35 kg/m2
5. Normal uterine anatomy
6. Normal pap test and Human papillomavirus (HPV) negative
7. Negative infection screen (HIV, HepB, HepC, Syphilis, gonorrhea, chlamydia)
8. Received counseling regarding alternatives to uterus donation such as adoption and gestational surrogacy
9. Fluent in the English Language
10. Willing to comply with screening, protocol and all required procedures
11. Has adequate social support
12. Compatible blood type with recipient
13. Negative flow cytometric crossmatch with recipient
14. Has current health insurance
15. Able to stay in the Philadelphia region for 3 weeks following uterus donation

Living Donor Participant Exclusion Criteria:

1. Previous multiple major abdominal/pelvic surgery
2. Severe endometriosis
3. History of hypertension, diabetes mellitus, thrombophilia or other clotting or bleeding disorders, significant heart, liver, kidney or central nervous system disease
4. History or obvious evidence of previous multiple/significant uterine surgery. Defined as >1 cesarean delivery and/or myomectomy
5. History of previous cervical surgery (cone biopsy or loop electrosurgical excision procedure)
6. Significant systemic disease (diabetes or systemic lupus erythematosus)
7. Previous obstetric problem including delivery <34 weeks and abnormal placental location (i.e. placenta Previa/accreta/increta/percreta)
8. Pregnancy
9. Abnormal uterine cavity
10. Vascular calcification on imaging tests
11. History of significant psychiatric illness
12. Current smoker (smoking cessation must have occurred 3 months prior to enrollment)
13. Chemical and/or alcohol dependency or abuse
14. Psychosocial problems (including alcoholism, drug abuse, documented behavioral disorders)
15. Unwilling to receive a transfusion of blood or blood products
16. Evidence of coercion or exchange of money or goods for donating the organ

Deceased Donor Inclusion Criteria:

1. Hemodynamically stable donor
2. Age between 18 to 50 years
3. Compatible blood type with recipient
4. Negative flow cytometric crossmatch with recipient
5. Live birth to miscarriage ratio ≥1
6. Normal gross uterine anatomy (as visually assessed by gynecologic surgeon at time of organ procurement)
7. Macroscopically normal cervix (polyp acceptable)
8. Negative infection screen (HIV, HepB, HepC, Syphilis)
9. Cytomegalovirus (CMV)- matched based on rapid donor screening. A CMV positive donor may be used in a CMV negative recipient. A CMV negative donor may be used in either a CMV positive or negative recipient.
10. Donates after brain death

Deceased Donor Exclusion Criteria:

1. Current malignancy or history of malignancy active within the past 5 years (Except adequately treated localized basal or squamous cell carcinoma of skin without evidence of recurrence)
2. No history or obvious evidence of previous multiple/significant uterine surgery. Defined as >1 cesarean delivery and/or myomectomy
3. No history or obvious evidence of previous cervical surgery (cone biopsy or loop electrosurgical excision procedure)
4. Significant systemic disease (i.e. diabetes, peripheral vascular or cardiovascular disease, autoimmune disease, renal or liver failure, etc.)
5. Previous obstetric problem including delivery <34 weeks and abnormal placental location (i.e. placenta Previa/accreta/increta/percreta)
6. Pregnancy
7. BMI >35 kg/m2
8. Donates after cardiac death (DCD)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female sex; specifically XX-bearing individual
Enrollment: 10 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Recipient: Successful engraftment of deceased or living donor uterus | Assessed 6 months after transplant
  Uterus remains in recipient with no complications (i.e. infection or rejection) or any complications that did arise could be successfully treated.
Recipient: Live-born child per embryo transfer | Assessed up to 35 weeks post-embryo transfer
Living Donor: Survival post-donation | Assessed at 2 years post-hysterectomy
  Living or deceased

SECONDARY OUTCOMES:
Recipient: Neonatal growth | Assessed at birth
  Birth weight percentile at delivery
Recipient: Pregnancy complications | Assessed up to 35 weeks post-embryo transfer
  Including but not limited to preeclampsia, gestational hypertension, gestational diabetes, and cholestasis of pregnancy.
Recipient: Surgical or medical complications following cesarean delivery | Assessed up to 6 months after delivery
Recipient: Surgical or medical complications following hysterectomy | Assessed 2 years after hysterectomy
Recipient: Child height percentile | Assessed at 2 years
Recipient: Child weight percentile | Assessed at 2 years
Living Donor: Intraoperative/postoperative/pregnancy/postpartum complications | Assessed at 2 years post-hysterectomy
Living Donor: Symptomatic claudication of buttock or legs | Assessed at 2 years post-hysterectomy
  yes or no
Living Donor: Genitourinary tract complications | Assessed at 2 years post-hysterectomy
Living Donor: Need for reoperation | Assessed at 2 years post-hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E O'Neill, MD, MTR, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Select trial data may be shared with the International Society of Uterine Transplantation (ISUTx) Registry. No protected health information will be shared.

REFERENCES:
- [Background] Griffin JE, Edwards C, Madden JD, Harrod MJ, Wilson JD. Congenital absence of the vagina. The Mayer-Rokitansky-Kuster-Hauser syndrome. Ann Intern Med. 1976 Aug;85(2):224-36. doi: 10.7326/0003-4819-85-2-224. PMID 782313
- [Background] White PM. "One for Sorrow, Two for Joy?": American embryo transfer guideline recommendations, practices, and outcomes for gestational surrogate patients. J Assist Reprod Genet. 2017 Apr;34(4):431-443. doi: 10.1007/s10815-017-0885-7. Epub 2017 Feb 9. PMID 28185120
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Consideration of the gestational carrier: a committee opinion. Fertil Steril. 2013 Jun;99(7):1838-41. doi: 10.1016/j.fertnstert.2013.02.042. Epub 2013 Mar 29. PMID 23541404
- [Background] Drabiak K, Wegner C, Fredland V, Helft PR. Ethics, law, and commercial surrogacy: a call for uniformity. J Law Med Ethics. 2007 Summer;35(2):300-9. doi: 10.1111/j.1748-720X.2007.00139.x. PMID 17518856
- [Background] O'Leary JA, Feldman M, Gaensslen DM. Uterine and tubal transplantation. Fertil Steril. 1969 Sep-Oct;20(5):757-60. doi: 10.1016/s0015-0282(16)37148-5. No abstract available. PMID 5822860
- [Result] Brannstrom M, Bokstrom H, Dahm-Kahler P, Diaz-Garcia C, Ekberg J, Enskog A, Hagberg H, Johannesson L, Kvarnstrom N, Molne J, Olausson M, Olofsson JI, Rodriguez-Wallberg K. One uterus bridging three generations: first live birth after mother-to-daughter uterus transplantation. Fertil Steril. 2016 Aug;106(2):261-6. doi: 10.1016/j.fertnstert.2016.04.001. Epub 2016 Apr 25. PMID 27125227
- [Result] Nair A, Stega J, Smith JR, Del Priore G. Uterus transplant: evidence and ethics. Ann N Y Acad Sci. 2008 Apr;1127:83-91. doi: 10.1196/annals.1434.003. PMID 18443334
- [Result] McKay DB, Josephson MA. Pregnancy in recipients of solid organs--effects on mother and child. N Engl J Med. 2006 Mar 23;354(12):1281-93. doi: 10.1056/NEJMra050431. No abstract available. PMID 16554530
- [Result] Saso S, Clarke A, Bracewell-Milnes T, Saso A, Al-Memar M, Thum MY, Yazbek J, Del Priore G, Hardiman P, Ghaem-Maghami S, Smith JR. Psychological Issues Associated With Absolute Uterine Factor Infertility and Attitudes of Patients Toward Uterine Transplantation. Prog Transplant. 2016 Mar;26(1):28-39. doi: 10.1177/1526924816634840. PMID 27136247
- [Result] Brannstrom M. Uterus transplantation and beyond. J Mater Sci Mater Med. 2017 May;28(5):70. doi: 10.1007/s10856-017-5872-0. Epub 2017 Mar 29. PMID 28357688
- [Result] Flyckt RL, Farrell RM, Perni UC, Tzakis AG, Falcone T. Deceased Donor Uterine Transplantation: Innovation and Adaptation. Obstet Gynecol. 2016 Oct;128(4):837-842. doi: 10.1097/AOG.0000000000001617. PMID 27607877
- [Result] Testa G, Koon EC, Johannesson L, McKenna GJ, Anthony T, Klintmalm GB, Gunby RT, Warren AM, Putman JM, dePrisco G, Mitchell JM, Wallis K, Olausson M. Living Donor Uterus Transplantation: A Single Center's Observations and Lessons Learned From Early Setbacks to Technical Success. Am J Transplant. 2017 Nov;17(11):2901-2910. doi: 10.1111/ajt.14326. Epub 2017 May 23. PMID 28432742
- [Derived] Johannesson L, Humphries LA, Porrett PM, Testa G, Anderson S, Walter JR, Rush M, Ferrando CA, O'Neill K, Richards EG. Classification and treatment of vaginal strictures at the donor-recipient anastomosis after uterus transplant. Fertil Steril. 2024 Sep;122(3):525-534. doi: 10.1016/j.fertnstert.2024.04.019. Epub 2024 Apr 16. PMID 38636770
- [Derived] Walter JR, Johannesson L, Falcone T, Putnam JM, Testa G, Richards EG, O'Neill KE. In vitro fertilization practice in patients with absolute uterine factor undergoing uterus transplant in the United States. Fertil Steril. 2024 Sep;122(3):397-405. doi: 10.1016/j.fertnstert.2024.04.017. Epub 2024 Apr 15. PMID 38631504
- See also: Please visit the UPENN Study Web Page — https://clinicalresearch.itmat.upenn.edu/clinicaltrial/4821/congenital-abnormalitiesfemale-infertility-penn-ut/